CLINICAL TRIAL: NCT03803995
Title: Mapping and Pacing of the His Bundle for Heart Failure Patients With Left Bundle Branch Block
Acronym: MAP HIS HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD 969
Record Dates: First submitted 2019-01-04; First posted 2019-01-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Left Bundle-Branch Block
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mapping and Pacing the His Bundle (Other): All patients will be in this arm. Mapping and Pacing the His Bundle will be performed.
  Interventions: Procedure: Mapping and Pacing the His Bundle; Procedure: Placing a guidewire in Coronary sinus for measurement of Q-LV during His Bundle pacing or, if needed, for LV pacing

INTERVENTIONS:
Procedure: Mapping and Pacing the His Bundle — During the device implant procedure, 3D electro-anatomical mapping of the His Bundle region will be performed using EnSite™ Precision™ mapping system and Advisor™ HD Grid mapping catheter. This procedure might be part of the standard-of-care at the participating centers.
Procedure: Placing a guidewire in Coronary sinus for measurement of Q-LV during His Bundle pacing or, if needed, for LV pacing — During the device implant procedure, a VisionWire coronary guidewire will also be placed into a branch of coronary sinus (CS), targeting a lateral branch. This guidewire could be used for collecting local left ventricle (LV) activation time (Q-LV) or pacing the LV. This guidewire could also be used to deliver a LV lead at physician's discretion. This procedure might be part of the standard-of-care at the participating centers.

SUMMARY:
This is a prospective, single-arm, non-randomized, non-blinded study designed to characterize the locations of His Bundle (HB) pacing that results in correction of electrical dyssynchrony and to characterize morphology and activation time of local intracardiac electrogram (IEGM) with an electro-anatomical mapping system during a device implant procedure and secondarily to assess the efficacy of HB pacing or HB plus LV pacing (when indicated) in correction of electrical dyssynchrony in heart failure patients with left bundle branch block.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are undergoing implant of an Abbott pacemaker or CRT device under standard indications
2. An ECG with a wide QRS complex (>130 ms)
3. ECG morphology of typical complete LBBB,
4. Patients have heart failure with NYHA Class II-IV symptoms,
5. LV EF <50%
6. At least 18 years old and not pregnant.
7. Must provide written informed consent prior to any clinical investigation related procedure.
8. Willing to comply with study evaluation requirements
9. Female subjects of child-bearing potential are required to have a negative pregnancy test done within 7 days prior to the implant procedure per site standard test. Female patients of childbearing potential should be instructed to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release.)

Exclusion Criteria:

1. Patients have non-specific intraventricular conduction delay or right bundle branch block
2. Previously implanted cardiac devices with three or more permanent leads
3. History of aortic valve repair or replacement
4. History of tricuspid valve replacement
5. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
6. Recent (< 3 months) myocardial infarction, ablation, electrolyte imbalance, or any condition within the last 90 days that would contraindicate for pacemaker or CRT implant in the opinion of the investigator
7. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Successful HB pacing sites | At device implant procedure
  Collect 3D Locations and electrogram characteristics (morphology and activation time) at the sites where His Bundle (HB) pacing is associated with left bundle recruitment and corrects electrical dyssynchrony at HB pacing implant procedure.

SECONDARY OUTCOMES:
Success rate of HB pacing | At device implant procedure
  Measure success rate of HB pacing or HB plus Left ventricular (LV) pacing in the correction of electrical dyssynchrony at implant procedure;
Ventricular activation during HB pacing | At device implant procedure
  Collect ventricular activation times during HB pacing or HB plus LV pacing as compared with intrinsic rhythm and other pacing configurations at implant procedure;
Echocardiographic measurements of LV ejection fraction | At three-month follow-up
  Collect echo measurements of LV ejection fraction at three-month follow-up visit
Echocardiographic measurements of LV end-systolic volume | At three-month follow-up
  Collect echo measurements of LV end-systolic volume at three-month follow-up visit
Capture threshold of HB pacing | Implant procedure, up to 3 days after implant procedure, two-week follow-up visit, three-month follow-up visit
  Measure capture threshold in volts of HB pacing at implant and at follow-up visits post implant
Lead impedance of HB pacing lead | Implant procedure, up to 3 days after implant procedure, two-week follow-up visit, three-month follow-up visit
  Measure lead impedance in ohms of HB pacing lead at implant and at follow-up visits post implant
Sensing amplitude of HB pacing lead | Implant procedure, up to 3 days after implant procedure, two-week follow-up visit, three-month follow-up visit
  Measure sensing amplitude in millivolts of HB pacing lead at implant and at follow-up visits post implant

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States